CLINICAL TRIAL: NCT05499325
Title: Requests for Medical Termination of Pregnancy for Psychological or Social Maternal Reasons at the "Maison Des Femmes" in Saint-Denis : Retrospective Study Between 2016 and 2022
Brief Title: Requests for Medical Termination of Pregnancy for Psychological or Social Maternal Reasons
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: CHSD_0028_MATER
Record Dates: First submitted 2022-08-11; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Pregnancy Related
Keywords: Medical termination of pregnancy; Psychic or social reason

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
When the request for termination of pregnancy is made at a term of less than sixteen weeks of amenorrhea, the patients have complete decision-making autonomy. This is called voluntary termination of pregnancy. On the other hand, when they are made after this term, their requests must be subject to a multidisciplinary assessment. This is called medical termination of pregnancy for maternal indication. Schematically, there are two categories of indications: "organic" (progressive cancer, severe heart disease, etc.) and "psycho-social". In the latter case, and although the recommendations of the CNGOF recommend a formalization of these requests in the centers where the patients are received, strong disparities are observed in practice. In addition, there are few epidemiological and clinical data concerning these medical terminations of pregnancy with a psychological or social maternal indication in the literature.

The objective of this work is to describe the demographic characteristics of patients who have made a request for termination of pregnancy after the legal deadline for psychological or social maternal reasons, and to specify the care pathways of these patients.

DETAILED DESCRIPTION:
Retrospective cohort (from 01/01/2016 to 02/28/2022) single-centre involving data from patients followed at the Maison des Femmes, and eligible for the study.

The demographic and care pathway variables will be the subject of a descriptive statistical analysis.

Expected results: improvement of knowledge relating to patients who consulted for termination of pregnancy after sixteen weeks of amenorrhea and their care pathway.

Outlook:

* Improving the knowledge of health professionals and therefore of care pathways, with a view to a more homogeneous use of legal systems.
* Improvement and simplification of care pathways.

ELIGIBILITY:
Inclusion Criteria:

* Minor or adult patients who have been seen at the Maison des Femmes in the context of a request for termination of pregnancy for psychological and/or social maternal reasons, including patients subject to a legal protection measure (guardianship , curators) during the consultation
* Consultation between 01/01/2016 and 02/28/2022

Exclusion Criteria:

* Refusal of inclusion in a study explained in the medical file (patient or guardian)
* Objection to the use of data or refusal to participate (patient or guardian)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients followed at the Maison des Femmes, having consulted between 01/01/2016 and 02/28/2022, having undergone a medical termination of pregnancy for psychological or social maternal reasons
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-08-17 (Estimated); Primary Completion 2022-08-17 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
age | Day 1
  epidemiology of patients who have undergone medical termination of pregnancy for psychological or social maternal reasons
place of life | Day 1
  epidemiology of patients who have undergone medical termination of pregnancy for psychological or social maternal reasons
social security | Day 1
  epidemiology of patients who have undergone medical termination of pregnancy for psychological or social maternal reasons
level of studies | Day 1
  epidemiology of patients who have undergone medical termination of pregnancy for psychological or social maternal reasons
occupation / resources | Day 1
  epidemiology of patients who have undergone medical termination of pregnancy for psychological or social maternal reasons
marital status | Day 1
  epidemiology of patients who have undergone medical termination of pregnancy for psychological or social maternal reasons
number of children | Day 1
  epidemiology of patients who have undergone medical termination of pregnancy for psychological or social maternal reasons
native country | Day 1
  epidemiology of patients who have undergone medical termination of pregnancy for psychological or social maternal reasons
recent life events | Day 1
  epidemiology of patients who have undergone medical termination of pregnancy for psychological or social maternal reasons

SECONDARY OUTCOMES:
migratory route | Day 1
  care pathway for patients who have undergone medical termination of pregnancy for psychological or social maternal reasons
medical and surgical history | Day 1
  care pathway for patients who have undergone medical termination of pregnancy for psychological or social maternal reasons
gynecological follow-up, and follow-up of the current pregnancy | Day 1
  care pathway for patients who have undergone medical termination of pregnancy for psychological or social maternal reasons

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital DELAFONTAINE, Saint-Denis, Île-de-France Region, France

REFERENCES:
- See also: Women victims of violence — https://www.lamaisondesfemmes.fr/jai-besoin-daide/nos-parcours-de-soins/